CLINICAL TRIAL: NCT07148934
Title: Validity and Algorithm Development for Detection of Supraventricular Tachycardia in Children-A Clinical Pilot Study
Status: Not yet recruiting | Type: Observational
Sponsor: University of Turku (Other)
Responsible Party: Principal Investigator, Anna Axelin, Professor, Head of Department, University of Turku
Other Study IDs: FIMEA/2025/002511-2
Record Dates: First submitted 2025-08-22; First posted 2025-08-29 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Supraventricular Tachycardia; Atrial Fibrillation (AF)
Keywords: Supraventricular Tachycardia; Atrial Fibrillation; Seismocardiography; SmartPhone
MeSH Terms: conditions — Tachycardia, Supraventricular; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study( SVT) Group: Children aged 0-10 years treated in the pediatric wards of Tyks Lighthouse Hospital with diagnosed or suspected supraventricular tachycardia (SVT).
  Interventions: Diagnostic Test: Smartphone seismographic recording and Bed Based Ballistocardiographic recordings
- Control Group: Children aged 0-10 years treated in the pediatric wards of Tyks Lighthouse hospital who have not been diagnosed with SVT (i.e., have a normal sinus rhythm).
  Interventions: Diagnostic Test: Smartphone seismographic recording and Bed Based Ballistocardiographic recordings

INTERVENTIONS:
Diagnostic Test: Smartphone seismographic recording and Bed Based Ballistocardiographic recordings — A short recording of heart rhythm using a smartphone and bed-based ballistocardiogram.

SUMMARY:
The aim of this study is to evaluate the reliability of smartphone seismocardiography (SCG) and bed-based ballistocardiography (BCG) for detecting supraventricular tachycardia (SVT) in children aged 0-10 years. The performance of these methods will be compared to the gold standard of continuous telemetry ECG recording.

DETAILED DESCRIPTION:
This study aims to validate the use of a cardiac monitoring system, comprising a smartphone for seismocardiography (SCG) and a smart mattress for ballistocardiography (BCG), to detect supraventricular tachycardia (SVT) in children aged 0-10 years. Additionally, the study will compare heart rate and breathing rate measurements from these investigational devices against a Philips Intellivue X2 ECG Monitor, which serves as the gold standard. A convenience sample of up to 60 children (30 in the SVT group and 30 in the control group) will be recruited, and their parents will also be interviewed to explore their perceptions of arrhythmia monitoring. The primary objective is to develop and understand algorithms for differentiating SVT from sinus rhythm using SCG and BCG signals.

ELIGIBILITY:
Inclusion Criteria:

* For children in Study(SVT) group:

  1. received informed consent from both parents/guardians
  2. the child is treated in the Pediatric wards of Tyks Lighthouse hospital
  3. the child is between the age of 0-10 years
  4. the child has diagnosed or suspected SVT.
* For children in control group:

  1. received informed consent from both parents/guardians
  2. the child is treated in the Pediatric wards of Tyks Lighthouse hospital
  3. the child is between the age of 0-10 years
  4. child has not diagnosed with SVT

Exclusion Criteria:

* All participant groups:

  1. not reaching the inclusion criteria

Ages: 0 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: N=up to 60, 30 for the study (SVT) group and 30 for the control group.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-12-15 (Estimated); Study Completion 2027-06-15 (Estimated)

PRIMARY OUTCOMES:
Algorithm development for Seismocardiograph and Ballistocardiograph for detecting Supraventricular tachycardia | 2025-2027
  Understanding and developing the algorithm to differentiate the supraventricular tachycardia (SVT) and sinus rhythm subjects based on seismocardiography and ballistocardiography signals.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Turku, Turku, Finland

IPD SHARING:
Plan to Share IPD: Undecided